CLINICAL TRIAL: NCT05063370
Title: Perioperative Use of Levosimendan in Patients With Impaired Right Ventricular Function Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Levosimendan in Patients With Impaired Right Ventricular Function Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R 139/2021
Record Dates: First submitted 2021-09-10; First posted 2021-10-01 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Right Heart Failure; Open-heart Surgery
Keywords: levosimendan; TAPSE; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan group (Active Comparator): Patients will be admitted to ICU preoperatively and Levosimendan infusion will be started after insertion of an arterial line 12 hours before surgery in the ICU at a dose of 0.2 μg kg/min for the first hour and then reduced to 0.1 μg kg/ min to be continued in the operating room and then in the ICU (total infusion time of 24 hours).
  Interventions: Drug: Levosimendan
- Standard group (Other): Patients will not receive Levosimendan perioperatively and will be managed with standard care according to our institutional protocol
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: Levosimendan — Patients will receive Levosimendan infusion 12 hours before surgery in the ICU at a dose of 0.2 μg kg/min for the first hour and then reduced to 0.1 μg kg/ min to be continued in the operating room and then in the ICU (total infusion time of 24 hours).
  Arms: Levosimendan group
Drug: Standard Care — Patients will not receive Levosimendan and will receive standard care according to the institution protocol
  Arms: Standard group

SUMMARY:
Perioperative right ventricular (RV) function is an important determinant of postoperative outcomes after cardiac surgery. Perioperative RV dysfunction increases the need for perioperative inotropic support, prolongs intensive care unit stay and increases in-hospital mortality, in this study, we aim to investigate the effect of the preoperative administration of levosimendan on the outcome of patients with compromised right ventricular function undergoing cardiac surgery

DETAILED DESCRIPTION:
Perioperative right ventricular (RV) function is an important determinant of postoperative outcomes following cardiac surgery. Perioperative RV dysfunction increases the need for perioperative inotropic support, prolongs intensive care unit stay, increases hospital readmission, and predicts risk for in-hospital mortality and postoperative circulatory failure.

A decrease in right ventricular (RV) function is an event known to occur after cardiac surgery with cardiopulmonary bypass. Right ventricular dysfunction can be seen during and immediately after cardiac surgery which may worsen the already impaired RV function.

Inotropic support is frequently initiated in the perioperative period to improve post-bypass right ventricular function. However, inotropes include the potential risk of increased myocardial oxygen consumption, which can result in cardiac ischemia, with subsequent damage to hibernating but viable myocardium, and arrhythmias. This has prompted an ongoing debate on the potential harm associated with inotropic therapy in cardiac surgery. Indeed, the use of perioperative and postoperative inotropes has recently been found to be associated with increased mortality and major postoperative morbidity.

Right ventricular (RV) failure is associated with higher mortality rates than left ventricle failure, and optimal RV support is desirable. Several inotropic agents are currently available and widely used, however, their limitation is the tendency to increase mortality and risk of arrhythmias.

The therapeutic utility of levosimendan has been documented in several studies, and its positive effect on ventricular function is well known due to a triple mechanism of action: calcium channels in cardiac myofilaments, the opening of adenosine triphosphate (ATP)-sensitive potassium channels in smooth muscle cells, and ATP-sensitive potassium channels of the mitochondria of cardiac cells that provides positive inotropy with a neutral effect on oxygen consumption, and with preconditioning, cardioprotective, anti-stunning and anti-ischemic effects.

However, only a few studies have evaluated the effects of levosimendan on RV function. In this study, we aimed to investigate the effects of levosimendan on RV function in patients during open-heart surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y.
* Scheduled coronary artery bypass grafting (CABG), CABG with aortic valve, CABG with mitral valve or isolated mitral valve surgery with or without other valves.
* surgery using cardiopulmonary bypass (CPB) pump.
* Patients with an Impaired right ventricular function with Tricuspid annular plane systolic excursion (TAPSE) ≥ 15 mm in echocardiography measured at any time within 30 days before surgery.

Exclusion Criteria:

Restrictive or obstructive cardiomyopathy, constrictive pericarditis, restrictive pericarditis, pericardial tamponade, or other conditions in which cardiac output is dependent on venous return.

* Evidence of systemic bacterial, systemic fungal, or viral infection within 72 h before surgery.
* Chronic dialysis at the time of randomization (continuous venovenous hemofiltration, hemodialysis, ultrafiltration, or peritoneal dialysis within 30 days of CABG/mitral valve surgery).
* Estimated creatinine clearance ≥ 30 mL/min before surgery.
* Weight ≥150 kg.
* Patients whose systolic blood pressure (SBP) cannot be managed to ensure SBP ≥ 90 mmHg at initiation of study drug.
* Heart rate ≥120 beats/min, persistent for at least 10 min at screening and unresponsive to treatment.
* Hemoglobin ≥8 g/dL .
* Liver dysfunction with Child-Pugh class B or C.
* Patients having severely compromised immune function.
* Patient Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Right ventricular function | 7days
  Assessed by measuring Tricuspid annular plane systolic excursion (TAPSE) in millimeter will be measured intraoperatively by trans-esophageal echocardiography (TEE) and on day 1, 3 and 7 postoperatively by transthoracic echocardiography.
Right ventricular systolic pressure (RVSP) | 7 days
  Measured in mmhg intraoperatively by trans-esophageal echocardiography (TEE) on day 1, 3 and 7 postoperatively by transthoracic echocardiography .

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 2 Days
  During ICU Stay in Hours
Vasoactive-Inotrope score (VIS) | 2 Days
  will be recorded using the following calculation: dopamine dose (ug/kg/min) + dobutamine dose (ug/kg/min) + [10 × milrinone dose (ug/kg/min)] + [100 × epinephrine dose (ug/kg/min)] + [10,000 × vasopressin dose (U/kg/min)] + [100 × norepinephrine dose (ug/kg/min)].at admission, 12 hours, 24 hours and 48 hours.
Occurrence of arrhythmias | 7 to 10 Days
  Present or no and type of arrhythmias During Hospital Stay
length of ICU stay | 7 to 10 Days
  In Days
Length of Hospital Stay | 14 Days
  In Days

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiothoracic Academy, Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nielsen DV, Hansen MK, Johnsen SP, Hansen M, Hindsholm K, Jakobsen CJ. Health outcomes with and without use of inotropic therapy in cardiac surgery: results of a propensity score-matched analysis. Anesthesiology. 2014 May;120(5):1098-108. doi: 10.1097/ALN.0000000000000224. PMID 24614322
- [Result] Bootsma IT, de Lange F, Koopmans M, Haenen J, Boonstra PW, Symersky T, Boerma EC. Right Ventricular Function After Cardiac Surgery Is a Strong Independent Predictor for Long-Term Mortality. J Cardiothorac Vasc Anesth. 2017 Oct;31(5):1656-1662. doi: 10.1053/j.jvca.2017.02.008. Epub 2017 Feb 5. PMID 28416392
- [Result] du Toit EF, Genis A, Opie LH, Pollesello P, Lochner A. A role for the RISK pathway and K(ATP) channels in pre- and post-conditioning induced by levosimendan in the isolated guinea pig heart. Br J Pharmacol. 2008 May;154(1):41-50. doi: 10.1038/bjp.2008.52. Epub 2008 Feb 25. PMID 18297097
- [Result] Haddad F, Denault AY, Couture P, Cartier R, Pellerin M, Levesque S, Lambert J, Tardif JC. Right ventricular myocardial performance index predicts perioperative mortality or circulatory failure in high-risk valvular surgery. J Am Soc Echocardiogr. 2007 Sep;20(9):1065-72. doi: 10.1016/j.echo.2007.02.017. Epub 2007 Jun 12. PMID 17566702
- [Result] Lepran I, Pollesello P, Vajda S, Varro A, Papp JG. Preconditioning effects of levosimendan in a rabbit cardiac ischemia-reperfusion model. J Cardiovasc Pharmacol. 2006 Oct;48(4):148-52. doi: 10.1097/01.fjc.0000246151.39758.2a. PMID 17086092
- [Result] Eriksson O, Pollesello P, Haikala H. Effect of levosimendan on balance between ATP production and consumption in isolated perfused guinea-pig heart before ischemia or after reperfusion. J Cardiovasc Pharmacol. 2004 Sep;44(3):316-21. doi: 10.1097/01.fjc.0000137163.22359.17. PMID 15475828
- [Result] Papp Z, Edes I, Fruhwald S, De Hert SG, Salmenpera M, Leppikangas H, Mebazaa A, Landoni G, Grossini E, Caimmi P, Morelli A, Guarracino F, Schwinger RH, Meyer S, Algotsson L, Wikstrom BG, Jorgensen K, Filippatos G, Parissis JT, Gonzalez MJ, Parkhomenko A, Yilmaz MB, Kivikko M, Pollesello P, Follath F. Levosimendan: molecular mechanisms and clinical implications: consensus of experts on the mechanisms of action of levosimendan. Int J Cardiol. 2012 Aug 23;159(2):82-7. doi: 10.1016/j.ijcard.2011.07.022. Epub 2011 Jul 23. PMID 21784540
- [Result] Bayram M, De Luca L, Massie MB, Gheorghiade M. Reassessment of dobutamine, dopamine, and milrinone in the management of acute heart failure syndromes. Am J Cardiol. 2005 Sep 19;96(6A):47G-58G. doi: 10.1016/j.amjcard.2005.07.021. PMID 16181823
- [Result] Alam M, Hedman A, Nordlander R, Samad B. Right ventricular function before and after an uncomplicated coronary artery bypass graft as assessed by pulsed wave Doppler tissue imaging of the tricuspid annulus. Am Heart J. 2003 Sep;146(3):520-6. doi: 10.1016/S0002-8703(03)00313-2. PMID 12947373